CLINICAL TRIAL: NCT01129401
Title: Evaluation of a Harm Reduction Treatment for Methamphetamine-Using Men Who Have Sex With Men (MSM)
Brief Title: Stonewall Treatment Evaluation Project
Acronym: STEP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: California HIV/AIDS Research Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR08-SF-423
Record Dates: First submitted 2010-05-06; First posted 2010-05-24 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Substance Abuse; HIV Infections
Keywords: methamphetamine; men who have sex with men; HIV/AIDS
MeSH Terms: conditions — Substance-Related Disorders; HIV Infections; Homosexuality; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stonewall Project Participants (Other)
  Interventions: Behavioral: Stonewall Project

INTERVENTIONS:
Behavioral: Stonewall Project — The Stonewall Project is an outpatient substance abuse treatment program for methamphetamine-using MSM that includes individual counseling, group counseling, and visits with a psychiatrists where indicated.

SUMMARY:
This treatment outcome evaluation of the Stonewall Project will recruit 150 participants to complete a face-to-face assessment visit at baseline, 3-month follow-up, and 6-month follow-up to examine treatment outcome with respect to HIV risk and substance use.

DETAILED DESCRIPTION:
Stonewall Project clients who have initiated treatment within the past 60 days will be eligible for the outcome evaluation. 20% of clients are likely to be on parole or probation; these clients will be eligible to participate in the study.

Outcome measures that will be examined as part of the treatment outcome evaluation include: 1) self-reported substance use; 2) urine toxicology screening; and 3) sex risk taking.

ELIGIBILITY:
Inclusion Criteria:

- Participants in the outcome evaluation must have initiated services at the Stonewall Project within the past 60 days.

Exclusion Criteria:

- Inability to provide informed consent as judged by the Co-PI's and study team.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
stimulant use (measured via self-report and urine toxicology screening) | 3 and 6 month follow-ups
  Participants will complete a self-report measure that assesses substance use during the past month. We will examine the total number of days that stimulants (cocaine, crack, or methamphetamine) were used during the past month. We will also conduct urine toxicology screening to determine whether participants test positive for cocaine or methamphetamine metabolites at each study visit. This is an objective measure of recent stimulant use (i.e., during the past 72 hours).

SECONDARY OUTCOMES:
sexual risk taking | 3 and 6 month follow-ups
  Sexual risk taking will be assessed using a measure that allows our team to examine risk as a function of HIV status, partner type (i.e., insertive or receptive), and whether the participant was under the influence of methamphetamine. Sex risk for HIV-negative men will be defined as any unprotected anal intercourse, irrespective of the HIV serostatus of sex partners. Sex risk for HIV-positive men will be defined as unprotected anal intercourse with HIV-negative or unknown serostatus partners.

CONTACTS AND LOCATIONS:
Overall Officials: Adam W Carrico, Ph.D., Principal Investigator — University of California, San Francisco; William J Woods, Ph.D., Principal Investigator — University of California, San Francisco; Michael D. Siever, Ph.D., Principal Investigator — San Francisco AIDS Foundation
Locations (2):
- United States (2):
  - San Francisco AIDS Foundation, San Francisco, California
  - University of California, San Francisco, San Francisco, California

REFERENCES:
- See also: Related Info — http://www.stonewallsf.org/